CLINICAL TRIAL: NCT00111449
Title: A Phase 3 Multicenter Study to Assess the Efficacy and Safety of Etanercept 50 mg Twice Weekly in Psoriasis
Brief Title: Evaluating the Safety of Etanercept 50 mg Twice Weekly in Subjects With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030117
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Psoriasis
Keywords: Psoriasis, adults; skin, Phase 3; clinical trial, Amgen; etanercept, Enbrel®; moderate, severe
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to determine the effect of etanercept 50 mg twice weekly compared to placebo over 12 weeks on the psoriasis area and severity index (PASI) in subjects with psoriasis. This study will also evaluate the safety and tolerability of etanercept 50 mg twice weekly; determine the effect of etanercept 50 mg twice weekly on patient reported outcomes (PRO); and characterize the pharmacokinetics (PK) profile of etanercept 50 mg twice weekly.

ELIGIBILITY:
Inclusion Criteria: - Active, but clinically stable, plaque psoriasis involving greater than or equal to 10% of the body surface area - A minimum PASI score of 10 obtained during the screening period Exclusion Criteria: - Active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit - Evidence of skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of an investigational product on psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-06

PRIMARY OUTCOMES:
Achievement of 75% or greater improvement from baseline in the Psoriasis Area and Severity Index (PASI) after 12 weeks of double-blind treatment.

SECONDARY OUTCOMES:
Dermatology Live Quality Index (DLQI) response at week 12
Subject's assessment of itching and improvements from baseline in joint pain (visual analog scale [VAS]) at week 12
Psoriasis pain (VAS) at week 12
Functional Assessment of Chronic Illness Therapy (FACIT) fatigue scale at week 12
PASI 50, 75 and 90 response and improvement from baseline in PASI score during long-term therapy
Static physician's global assessment of psoriasis (sPGA) from baseline during long-term therapy
Adverse events, infections injection site reactions during long-term therapy
Serious adverse events and infections during long-term therapy
Clinical laboratory values, vital signs and antibodies to etanercept during long-term therapy

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Krishnan R, Cella D, Leonardi C, Papp K, Gottlieb AB, Dunn M, Chiou CF, Patel V, Jahreis A. Effects of etanercept therapy on fatigue and symptoms of depression in subjects treated for moderate to severe plaque psoriasis for up to 96 weeks. Br J Dermatol. 2007 Dec;157(6):1275-7. doi: 10.1111/j.1365-2133.2007.08205.x. Epub 2007 Oct 4. No abstract available. PMID 17916204
- [Result] Tyring S, Gottlieb A, Papp K, Gordon K, Leonardi C, Wang A, Lalla D, Woolley M, Jahreis A, Zitnik R, Cella D, Krishnan R. Etanercept and clinical outcomes, fatigue, and depression in psoriasis: double-blind placebo-controlled randomised phase III trial. Lancet. 2006 Jan 7;367(9504):29-35. doi: 10.1016/S0140-6736(05)67763-X. PMID 16399150
- [Result] Tyring S, Gordon KB, Poulin Y, Langley RG, Gottlieb AB, Dunn M, Jahreis A. Long-term safety and efficacy of 50 mg of etanercept twice weekly in patients with psoriasis. Arch Dermatol. 2007 Jun;143(6):719-26. doi: 10.1001/archderm.143.6.719. PMID 17576937
- [Derived] Papp K, Poulin Y, Vieira A, Shelton J, Poulin-Costello M. Disease characteristics in patients with and without psoriatic arthritis treated with etanercept. J Eur Acad Dermatol Venereol. 2014 May;28(5):581-9. doi: 10.1111/jdv.12138. Epub 2013 Mar 7. PMID 23465037
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20030117.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/